CLINICAL TRIAL: NCT05988918
Title: A Phase II Multicenter Trial of ESK981 in Patients With Select Solid Tumors
Brief Title: Multicenter Trial of ESK981 in Patients With Select Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2023.005; HUM00233810 (Other: University of Michigan)
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Adenocarcinoma; Adenosquamous Carcinoma; Pancreatic Neuroendocrine Tumor; Pancreatic Neuroendocrine Carcinoma; Gastrointestinal Neuroendocrine Tumor; Gastrointestinal Neuroendocrine Carcinoma; Neuroendocrine Prostate Carcinoma
MeSH Terms: conditions — Carcinoma, Adenosquamous; Adenoma, Islet Cell; Somatostatinoma; Gastro-enteropancreatic neuroendocrine tumor | interventions — 11-(2-methylpropyl)-12,13-dihydro-2-methyl-8-(pyrimidin-2-ylamino)-4H-indazolo(5,4-a)pyrrolo(3,4-c)carbazol-4-one

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort 1 (Experimental): Pancreatic adenocarcinoma
  Interventions: Drug: ESK981
- Cohort 2 (Experimental): Pancreatic or gastrointestinal neuroendocrine neoplasms with Ki-67 > 20%
  Interventions: Drug: ESK981
- Cohort 3 (Experimental): Neuroendocrine prostate carcinoma with Ki-67 > 20%
  Interventions: Drug: ESK981

INTERVENTIONS:
Drug: ESK981 — 160 mg, PO, Once daily 5 days on and 2 days off
  Other Names: CEP-11981

SUMMARY:
This protocol will enroll patients with pancreatic adenocarcinoma and adenosquamous carcinoma (Cohort 1), gastrointestinal/pancreatic neuroendocrine neoplasms with Ki-67 > 20% (Cohort 2) and neuroendocrine prostate carcinoma (Cohort 3)). Each cohort will have its own interim analysis after enrollment of 10 patients.

Subjects will be given a one-month (28 day) supply of study drug (ESK981). Subjects will be instructed to take 4 capsules, with or without food, once per day for 5 consecutive calendar days, then take a drug holiday for 2 consecutive days before repeating the 5 days on-2 days off cycle in sets of 4 weeks or 28 calendar days. Subjects will be asked to keep a pill diary noting the date they take their study drug.

ELIGIBILITY:
Eligibility Criteria:

* Patients with histological or cytological confirmation of advanced cancer per specific cohort.

  * Cohort 1: Pancreatic adenocarcinoma or adenosquamous carcinoma who have progressed or deemed intolerant of the standard of care chemotherapy regimens.
  * Cohort 2: Pancreatic or gastrointestinal neuroendocrine tumor or carcinoma with Ki-67 > 20% who have progressed or deemed intolerant of at least first-line standard of care systemic therapy.
  * Cohort 3: The subject has histologically proven prostate cancer who have progressed or deemed intolerant of at least first-line standard of care systemic therapy with radiologic evidence of metastases and at least one of the following:

    * Small cell or neuroendocrine morphology on the basis of tissue sample.
    * Prostate adenocarcinoma with IHC staining for neuroendocrine markers (e.g., chromogranin and synaptophysin).
    * Presence of visceral metastases or high-volume disease (> 4 sites of metastases) with a PSA ≤ 5.
    * Serum chromogranin A level ≥ 5x upper limit of normal (ULN) and/or serum neuron specific enolase (NSE) ≥ 2x ULN.
    * Trans-differentiated carcinoma or poorly-differentiated carcinoma
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2
* Must be ≥ 18 years of age.
* Evaluable disease determined using guidelines of Response Evaluation Criteria in Solid Tumors (RECIST version 1.1)
* Ability to understand and willingness to sign IRB-approved informed consent.
* Willing to provide archived tissue, if available, from a previous diagnostic biopsy.
* Must be able to tolerate CT and/or MRI with contrast.
* At least 4 weeks from major surgery with resolution of any sequela to date of enrollment
* Laboratory values ≤2 weeks during screening must be:

  * Platelet count ≥ 75,000 cells/mm3
  * Absolute neutrophil count ≥ 1500 cells/mm3
  * Hemoglobin ≥ 9 g/dL
  * AST/ALT ≤ 3x upper limit of normal [ULN], or (≤ 5x ULN if liver metastasis present)
  * Bilirubin ≤ 1.5x ULN, or (≤ 2.5 x ULN for subjects with Gilbert's syndrome)
  * Albumin ≥ 3 g/dL
  * Serum creatinine clearance CrCl ≥ 50 mL/min per Cockcroft-Gault Formula
  * INR ≤ 1.5 (or <2.0 if on anticoagulants)
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must agree to use acceptable highly effective contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive(s), intrauterine hormone releasing system (IUS), bilateral tubal occlusion or vasectomized partner) during and for 9 months after last study dose and must have a negative serum or urine pregnancy test during screening.
* Males with female partners (of childbearing potential) and female partners (of childbearing potential) with male partners must agree to use double barrier contraceptive measure (a combination of male condom with either cap, diaphragm or sponge with spermicide) in addition to oral contraception, or avoidance of intercourse during the study and for 6 months after last study dose is received.
* Female patients must not be pregnant, have a positive pregnancy test, breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 9 months after the last dose of study treatment.
* Male patients must be willing to abstain from donating sperm during treatment and for 6 months after completion of study treatment.
* No evidence of active infection and no serious infection within the past 30 days. Patient must have completed antibiotic course.
* No known cerebral metastasis, central nervous system (CNS), or epidural tumor (unless previously treated, asymptomatic and stable for at least 3 months).
* No active heart disease including but not limited to myocardial infarction that is <3 months prior to registration, symptomatic congestive heart failure (NYHA class 3 or 4), symptomatic coronary artery disease, symptomatic angina pectoris.
* No history of acute cerebrovascular disease, arterial or venous thromboembolism, percutaneous angioplasty, or coronary artery bypass surgery within 6 months prior to registration
* No pre-existing coagulopathy, or serious bleeding within 3 months prior to registration.
* No prior malignancy except for the following: adequately treated basal or squamous cell skin cancer, in situ cancer, localized prostate cancer (Gleason score <8), or adequately treated cancer from which the patient has been disease-free for at least 3 years prior to registration.
* Must not have uncontrolled diarrhea at the time of enrollment.
* Patients must not use a chronic daily medication known to be a strong or moderate inhibitor of CYP1A2, CYP2C8 or CYP3A4 at registration (as per Appendix II).
* Patients must have recovered to baseline or ≤ grade 1 CTCAE v5.0 from toxicities related to any prior treatments, unless adverse event(s) is deemed clinically non-significant and/or stable on supportive therapy.
* Patients must not have uncontrolled hypertension defined as blood pressure >150/90 despite optimal medical management.
* No known hypersensitivity to gelatin or lactose monohydrate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 4 months after initiating study drug
  Determining efficacy using proportion of patients alive and progression-free at 4 months within each cancer subtype

SECONDARY OUTCOMES:
Overall Response Rate (ORR) within each cancer subtype | up to 18 months from treatment discontinuation
  The ORR will be assessed per RECIST v1.1 criteria (Cohort 1 and 2) or combined RECIST v1.1 + PCWG3 criteria (Cohort 3). Partial or complete response will require confirmation on repeat scan at least 4 weeks from initial radiologic response
Duration of Response (DoR) within each cancer subtype | up to 18 months from treatment discontinuation
  DoR will be measured from the start date of the best response achieved until the date of relapse (i.e., progression). Continuing responders will be right-censored as of the most recent date on which their response status had been assessed. DoR applies to only the patients who achieve either a complete response or a partial response.
Overall Survival (OS) within each cancer subtype | up to 18 months from treatment discontinuation
  The OS will be defined from the date of treatment to either date of death or censoring and estimated using the product-limit method of Kaplan and Meier. Follow-up time will be censored at the date of last disease evaluation.
Safety and tolerability in each cancer subtype | up to 30 days from treatment discontinuation
  Adverse events (AEs) will be defined per the NCI Common Toxicity Criteria for Adverse Events (CTCAE) v5.0.
Median Progression- Free Survival (PFS) within each cancer subtype | up to 18 months from treatment discontinuation
  The PFS will be defined as time from date of initial treatment to date of radiological or clinical progression (leading to withdrawal from the study treatment), or death from any cause on study treatment, whichever comes first. Follow-up time will be censored at the date of last disease evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Vaibhav Sahai, Principal Investigator — University of Michigan
Locations (3):
- United States (3):
  - Rogel Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No